CLINICAL TRIAL: NCT00547040
Title: Arterial Stiffness and Calcifications in Incident Renal Transplant Recipients
Acronym: ASCIT
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kathleen Claes, md, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML3775
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2011-10

CONDITIONS: Renal Transplant; Atherosclerosis; Arterial Stiffness
Keywords: calcification; bone lesions
MeSH Terms: conditions — Atherosclerosis; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: incident renal transplant patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of this study is to determine the:

* Natural history of calcification posttransplantation
* Natural history of BMC following renal transplantation
* Reverse correlation between calcification score and aortic calcifications following renal transplantation
* Correlation of IMT, BMC, PWV and biochemical variables
* Correlation of IMT, BMC, PWV, biochemical variables and outcome
* Predictors of CV disease after transplantation
* Predictors of IMT progression, BMC loss and PWV progression after renal transplantation

ELIGIBILITY:
Inclusion Criteria:

* Incident renal transplant patients or combined renal/pancreas transplant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: incident renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
cardiovascular outcome | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: kathleen Claes, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Jorgensen HS, Claes K, Smout D, Naesens M, Kuypers D, D'Haese P, Cavalier E, Evenepoel P. Associations of Changes in Bone Turnover Markers with Change in Bone Mineral Density in Kidney Transplant Patients. Clin J Am Soc Nephrol. 2024 Apr 1;19(4):483-493. doi: 10.2215/CJN.0000000000000368. Epub 2023 Nov 29. PMID 38030558
- [Derived] Evenepoel P, Claes K, Viaene L, Bammens B, Meijers B, Naesens M, Sprangers B, Kuypers D. Decreased Circulating Sclerostin Levels in Renal Transplant Recipients With Persistent Hyperparathyroidism. Transplantation. 2016 Oct;100(10):2188-93. doi: 10.1097/TP.0000000000001311. PMID 27379556
- [Derived] Claes KJ, Heye S, Bammens B, Kuypers DR, Meijers B, Naesens M, Vanrenterghem Y, Evenepoel P. Aortic calcifications and arterial stiffness as predictors of cardiovascular events in incident renal transplant recipients. Transpl Int. 2013 Oct;26(10):973-81. doi: 10.1111/tri.12151. Epub 2013 Jul 19. PMID 23870026